CLINICAL TRIAL: NCT03654768
Title: A Randomized Phase II Study of Ruxolitinib (NSC-752295) in Combination With BCR-ABL Tyrosine Kinase Inhibitors in Chronic Myeloid Leukemia (CML) Patients With Molecular Evidence of Disease
Brief Title: Testing the Addition of Ruxolitinib to the Usual Treatment (Tyrosine Kinase Inhibitors) for Chronic Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1712; NCI-2017-02066 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1712 (Other: SWOG); S1712 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — bosutinib; Dasatinib; nilotinib; ruxolitinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (bosutinib, dasatinib, nilotinib, imatinib) (Active Comparator): Patients receive bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosutinib; Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Drug: Nilotinib; Drug: Imatinib
- Arm II (ruxolitinib phosphate, dasatinib, nilotinib, imatinib) (Experimental): Patients receive ruxolitinib phosphate PO BID on days 1-90, and bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Drug: Nilotinib; Drug: Ruxolitinib; Drug: Imatinib

INTERVENTIONS:
Drug: Bosutinib — Given PO
  Other Names: Bosulif; SKI 606; SKI-606
  Arms: Arm I (bosutinib, dasatinib, nilotinib, imatinib)
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nilotinib — Given PO
  Other Names: AMN107; NILOTINIB HYDROCHLORIDE MONOHYDRATE; Nilotinib Monohydrochloride Monohydrate; Tasigna
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Jakafi; Oral JAK Inhibitor INCB18424
  Arms: Arm II (ruxolitinib phosphate, dasatinib, nilotinib, imatinib)
Drug: Imatinib — Given PO
  Other Names: Gleevec®; STI-571

SUMMARY:
This randomized phase II trial studies how well ruxolitinib phosphate, and bosutnib, dasatinib, imatinib or nilotinib, work in treating patients with chronic myeloid leukemia. Chronic myeloid leukemia cells produce a protein called BCR-ABL. The BCR-ABL protein helps chronic myeloid leukemia cells to grow and divide. Tyrosine kinase inhibitors, such as bosutinib, dasatinib, and nilotinib, stop the BCR-ABL protein from working, which helps to reduce the amount of chronic myeloid leukemia cells in the body. Ruxolitinib is a different type of drug that helps to stop the body from making substances called growth factors. Chronic myeloid leukemia cells need growth factors to grow and divide. The addition of ruxolitinib to the tyrosine kinase inhibitor may or may not help reduce the amount of chronic myeloid leukemia cells in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the rate of molecular response 4.5 (MR4.5) after 12 months of combination therapy with ruxolitinib phosphate (ruxolitinib) plus a tyrosine-kinase inhibitor (TKI) (bosutinib, dasatinib, imatinib or nilotinib) versus a TKI alone, based on local polymerase chain reaction (PCR) testing to measure BCR-ABL transcripts in chronic phase chronic myelogenous leukemia (CML) patients with molecular evidence of disease.

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities of each regimen in this patient population.

II. To estimate progression free survival and overall survival of each regimen in this patient population.

ADDITIONAL OBJECTIVES:

I. To describe patterns of MR4.5 and molecular response 4.0 (MR4.0) attainment and failure over the 3, 6, 9, and 12-month time points of each regimen in this patient population.

II. To evaluate drug compliance based on patient reported drug intake calendars in this patient population.

III. To describe the kinetics of response in this patient population (as measured by quantitative BCR-ABL/BCR ratio) in both arms over the 3, 6, 9, and 12-month time points.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive bosutinib orally (PO) daily or dasatinib PO daily or nilotinib PO twice daily (BID) or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive ruxolitinib phosphate PO BID on days 1-90, and bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years, and then annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of chronic phase chronic myeloid leukemia without any history of progression to accelerated or blast phase CML; no new bone marrow aspiration and biopsy is needed to prove diagnosis prior to randomization; however, documentation stating the patient is in chronic phase is required
* Patients must have detectable BCR-ABL transcripts measured by reverse transcriptase (RT)-PCR at a clinical laboratory improvement act (CLIA)-approved laboratory and reported on the international scale (IS) with a value of > 0.0032% IS and =< 1.0% IS within 21 days prior to randomization; the RT-PCR assay must have the sensitivity to detect a 4.5 log reduction in BCR-ABL transcripts from 100% IS (0.0032% IS or lower)
* Patients must have been receiving TKI treatment for CML for at least 12 months prior to randomization. Hydroxyurea prior to initiation of TKI is allowed.
* Patients must be currently receiving treatment with bosutinib (within the allowable dose range of 200-500 mg daily), nilotinib (within the allowable dose range of 150-400 mg BID or a cumulative daily dose of 300-800 mg), dasatinib (within the allowable dose range of 40-140 mg daily), or imatinib (within the allowable dose range of 300-400 mg daily); they must have received their current TKI for a minimum of 6 months prior to randomization and must be expected to remain on the same TKI for the next 12 months
* Patient must not have a history of resistance to any prior TKI drug; if patient has received more than one TKI, the reason for changing treatment must have been something other than resistance or inadequate response to the prior TKI (for example, intolerance to the prior TKI) and the treatment change must have occurred >= 6 months prior to randomization.
* Patients must not be receiving any other investigational agents
* Patients must have complete history and physical examination within 28 days prior to randomization
* If clinically indicated, patients must have corrected Fridericia's correction formula (QTcF) interval < 500 ms (by Fridericia calculation) on a 12-lead electrocardiography (EKG) within 7 days prior to randomization
* Platelets >= 100,000/mm^3 (100.0 x 10^9/L) within 7 days prior to randomization
* Absolute neutrophil count (ANC) > 1,000/mm^3 (1.0 x 10^9/L) within 7 days prior to randomization
* Hemoglobin >= 8 g/dL within 7 days prior to randomization
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x institutional upper limit of normal (IULN) within 7 days prior to randomization
* Total bilirubin =< 1.5 x IULN within 7 days prior to randomization (unless the patient has a known diagnosis of Gilbert's syndrome)
* Serum creatinine =< 1.5 x IULN within 7 days prior to randomization
* Prior malignancy is allowed providing it does not require concurrent therapy; exception: active hormonal therapy is allowed
* Patients must not be pregnant or nursing due to the teratogenic potential of the drugs used on this study; women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to randomization; women/men of reproductive potential must have agreed to use an effective contraceptive method during treatment and for 30 days after discontinuation of study drug; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients known to be human immunodeficiency virus positive (HIV+) are eligible provided they meet all other eligibility criteria and have undetectable HIV viral loads on their most recent viral load test which must have been performed in the last 6 months
* Specimens (peripheral blood) must be collected and submitted to a CLIA-approved laboratory, within 21 days prior to randomization; BCR-ABL transcripts must be measured using RT-PCR and results must be reported using the international scale; the RT-PCR assay must have the sensitivity to detect a 4.5 log reduction in BCR-ABL transcripts from 100% IS (must be able to detect 0.0032% IS or lower)
* Patients must be offered participation in submission of specimens for central BCR-ABL quantification and banking for future specimens; this submission is highly encouraged as an important protocol endpoint; with patient's consent, specimens must be collected and submitted, within 21 days prior to randomization
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2028-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra L Sweet, Principal Investigator — SWOG Cancer Research Network
Locations (541):
- United States (541):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Providence Queen of The Valley, Napa, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Island Urology-Hilo, Hilo, Hawaii
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mercy Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Zhao H, Deininger M. Eradicating residual chronic myeloid leukaemia: basic research lost in translation. Lancet Haematol. 2021 Feb;8(2):e101-e104. doi: 10.1016/S2352-3026(21)00001-6. No abstract available. PMID 33513367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 participants were assessed for eligibility, 6 were ineligible (3 had no bone marrow at diagnosis, 2 had TKI switch due to resistance, and 1 was on TKI for less than a year). 75 participants were randomized, 38 to the Single Agent TKI arm and 37 to the TKI + Ruxolitinib arm.
Groups:
- Single Agent TKI: Patients receive bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
- TKI + Ruxolitinib: Patients receive ruxolitinib phosphate PO BID on days 1-90, and bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Started | 38 | 37
Completed | 33 | 22
Not Completed | 5 | 15
Not completed — Adverse Event | 1 | 6
Not completed — Loss of response | 2 | 2
Not completed — Non-compliance | 0 | 1
Not completed — Refusal not related to toxicity | 1 | 5
Not completed — Did not receive protocol therapy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Agent TKI | TKI + Ruxolitinib | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Median (Full Range); unit: years] | 55 [19 to 80] | 47 [20 to 78] | 50 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 29 | 21 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 24 | 29 | 53
  Unknown or Not Reported | 10 | 7 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 1 | 1 | 2
  Race: Pacific Islander | 1 | 0 | 1
  Race: Asian | 0 | 1 | 1
  Race: White | 33 | 29 | 62
  Race: Unknown | 3 | 6 | 9
ECOG PS [Count of Participants; unit: Participants] — ECOG Performance Status Scale range from 0 to 2, with higher scores reflecting greater disability.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    PS 0 | 26 | 25 | 51
    PS 1 | 12 | 11 | 23
    PS 2 | 0 | 1 | 1
Length on TKI [Count of Participants; unit: Participants]
  TKI: 1-4 years | 24 | 21 | 45
  TKI: 4-10 years | 14 | 16 | 30
TKI and Randomization [Count of Participants; unit: Participants]
  Bosutinib | 4 | 4 | 8
  Dasatinib | 22 | 24 | 46
  Imatinib | 5 | 2 | 7
  Nilotinib | 7 | 7 | 14
Molecular Response at Randomization [Count of Participants; unit: Participants] — Molecular Response was reported using the International Scale (IS)
  MMR: On the International Scale, this response is equivalent to a value of ≤0.1%.
  MR20: On the International Scale, this response is equivalent to a value of ≤1%.
  MR40: The patients BCR-ABL/BCR ratio must be at least 10,000 times (4.0 logs) smaller than100% IS , i.e., must demonstrate a 4.0-log reduction relative to100% IS. When reported on the International Scale, this response is equivalent to a value of ≤ 0.01%.
  Participants
    MMR | 21 | 20 | 41
    MR20 | 14 | 11 | 25
    MR40 | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Rate of Molecular Response 4.5 (MR4.5)
Description: The participants BCR-ABL/BCR ratio must be at least 31,623 times (4.5 logs) smaller than100% IS, i.e., must demonstrate a 4.5-log reduction relative to 100% IS. When reported on the International Scale (IS), this response is equivalent to a value of ≤ 0.0032%. Values are reported as percentages with a higher rate being better then a lower rate.
Time Frame: At 12 months
Population: This population includes the 75 eligible and evaluable participants. 38 in the Single Agent TKI arm and 37 in the TKI + Ruxolitnib arm.
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Number analyzed (Participants) | 38 | 37
percentage of participants | 3 | 14
Statistical Analysis 1: Comparison: Single Agent TKI vs TKI + Ruxolitinib; Test type: Superiority; p = 0.09, Fisher Exact

2. Secondary Outcome: Overall Survival
Description: Overall survival will be measured for all patients from the date of randomization until death from any cause with observations censored at the date of last contact for patients last known to be alive. The results were presented as 3-year OS estimate.
Time Frame: From the date of randomization until death from any cause with observations censored at the date of last contact for patients last known to be alive, assessed up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Number analyzed (Participants) | 38 | 37
percentage of participants | 100 [NA to NA] — Kaplan-Meier confidence intervals could not be estimated for the TKI alone arm because there were no events on that arm | 97 [80 to 100]
Statistical Analysis 1: Comparison: Single Agent TKI vs TKI + Ruxolitinib; Test type: Superiority; p = 0.30, Log Rank

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is measured from the date of randomization on study until the first of treatment failure/loss of response, progression, or death from any cause. Observations are censored at the date of last follow-up for patients last known to be alive without report of treatment failure/loss of response or progression.
Time Frame: From the date of randomization on study until the first of treatment failure/loss of response, progression, or death from any cause, assessed up to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Number analyzed (Participants) | 38 | 37
percentage of participants | 89 [74 to 96] | 89 [73 to 96]
Statistical Analysis 1: Comparison: Single Agent TKI vs TKI + Ruxolitinib; Test type: Superiority; p = 0.90, Log Rank

4. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. CTCAE Version 5.0 was used for all AE reporting.
Time Frame: Duration of treatment and follow-up until death or 5 years post registration.
Population: Participants who were eligible and received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Number analyzed (Participants) | 37 | 36
Participants
  Constipation | 0 | 1
  Fatigue | 0 | 1
  Headache | 0 | 1
  Hypertension | 1 | 0
  Nausea | 0 | 1
  Neutrophil count decreased | 1 | 2
  Pancreatitis | 1 | 0
  Pericardial effusion | 1 | 0
  Respiratory failure | 0 | 1
  Vomiting | 0 | 1

5. Secondary Outcome: MR4.5 Attainment
Description: Will be summarized descriptively
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Number analyzed (Participants) | 38 | 37
percentage of participants
  3-Month Response | 3 | 8
  6-Month Response | 3 | 5
  9-Month Response | 0 | 14
  12-Month Response | 3 | 14

6. Secondary Outcome: Molecular Rate 4.0 (MR 4.0) Attainment
Description: Will be summarized descriptively
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Number analyzed (Participants) | 38 | 37
percentage of participants
  3-Month Response | 16 | 24
  6-Month Response | 13 | 24
  9-Month Response | 18 | 22
  12-Month Response | 11 | 19

7. Secondary Outcome: Drug Compliance
Description: Will be summarized descriptively, results presented as number of participants that were fully compliant for all cycles that they received treatment.
Time Frame: Up to 5 years
Population: This population includes the 73 participants who were eligible and received at least one dose of study treatment. 37 in the Single Agent TKI arm and 36 in the TKI + Ruxolitnib arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
Number analyzed (Participants) | 37 | 36
Participants | 36 | 31

8. Secondary Outcome: BCR-ABL/BCR Comparison
Description: Quantitative RT-PCR measurement of BCR-ABL transcript levels on the International Scale (IS), expressed as log₁₀ ratios of BCR-ABL to ABL. Mean and standard deviation of log₁₀ BCR-ABL (IS) are reported at 3, 6, 9, and 12 months for each treatment arm. Lower values represent deeper molecular response.
  This scale ranges from 0 to -5, with a more negative number corresponding to a better outcome.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log₁₀ BCR-ABL Ratio
Groups:
- TKI + Ruxolitnib: Patients receive ruxolitinib phosphate PO BID on days 1-90, and bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | Single Agent TKI | TKI + Ruxolitnib
Number analyzed (Participants) | 38 | 37
Log₁₀ BCR-ABL Ratio
  3-months | -1.22 (0.52) | -1.37 (0.60)
  6-months | -1.30 (0.62) | -1.48 (0.64)
  9-months | -1.32 (0.60) | -1.47 (0.68)
  12-months | -1.26 (0.55) | -1.52 (0.68)

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 5 years post randomization.
Description: CTCAE version 5.0 was used for toxicity and SAEs reporting. There were 37 participants on the Single Agent TKI arm that were assessed for AEs, and 36 participants on the TKI + Ruxolitinib arm that were assessed for AEs.
Groups:
- Single Agent TKI: Patients receive bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. The number of participants at risk in All-cause Mortality are the number of participants who were randomized. The number of participants at risk in Serious Adverse Events are the number of participants who received at least one dose of protocol treatment.
- TKI + Ruxolitinib: Patients receive ruxolitinib phosphate PO BID on days 1-90, and bosutinib PO daily or dasatinib PO daily or nilotinib PO BID or imatinib PO daily on days 1-90. Treatment repeats every 90 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. The number of participants at risk in All-cause Mortality are the number of participants who were randomized. The number of participants at risk in Serious Adverse Events are the number of participants who received at least one dose of protocol treatment.
Arm/Group | Single Agent TKI | TKI + Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 0/38 | 1/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 4/36
Other Adverse Events (participants affected / at risk) | 31/37 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent TKI (N=37) | TKI + Ruxolitinib (N=36)
Fatigue (General disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent TKI (N=37) | TKI + Ruxolitinib (N=36)
Anemia (Blood and lymphatic system disorders) | 5 | 15
Palpitations (Cardiac disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 5 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 13
Dry mouth (Gastrointestinal disorders) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 16
Vomiting (Gastrointestinal disorders) | 3 | 5
Chills (General disorders) | 0 | 4
Edema limbs (General disorders) | 2 | 2
Fatigue (General disorders) | 9 | 18
Flu like symptoms (General disorders) | 1 | 2
General disorders and administration site conditio (General disorders) | 1 | 2
Infections and infestations-Other (Infections and infestations) | 3 | 3
Upper respiratory infection (Infections and infestations) | 2 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 2
Injury, poisoning and procedural complications-Oth (Injury, poisoning and procedural complications) | 0 | 3
Alanine aminotransferase increased (Investigations) | 4 | 10
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 12
Blood bilirubin increased (Investigations) | 1 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 2
Cholesterol high (Investigations) | 0 | 4
Creatinine increased (Investigations) | 5 | 6
Investigations-Other (Investigations) | 2 | 1
Lipase increased (Investigations) | 2 | 4
Lymphocyte count decreased (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 1 | 6
Platelet count decreased (Investigations) | 1 | 2
Weight gain (Investigations) | 1 | 3
Weight loss (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 2 | 7
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 4
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 9
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 3 | 8
Anxiety (Psychiatric disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 3 | 3
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 4
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03654768/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03654768/ICF_002.pdf